CLINICAL TRIAL: NCT01181960
Title: Research and Evaluation of Antipsychotic Treatment in Community Behavioral Health Organizations
Status: Completed | Type: Observational
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017107; RIS-OUT-239 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Risperidone long acting injectable; Risperdal Consta; Paliperidone Palmitate; Invega Sustenna
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 001: Risperidone long acting injectable - New Starts Patients who switch to Risperidone long acting injectable or receive an initial injection of Risperidone long acting injectable within the 30 days prior to enrollment will be eligible for inclusion in the Risperidone long acting injectable New Starts cohort.
  Interventions: Drug: Risperidone long acting injectable - New Starts
- 002: Risperidone long acting injectable - Continuous Users Patients who have been on Risperidone long acting injectable for at least 6 months before baseline with no gaps between injections of more than 30 days will be eligible for inclusion in the Risperidone long acting injectable Continuous Users cohort.
  Interventions: Drug: Risperidone long acting injectable - Continuous Users
- 003: Paliperidone Palmitate -New and Continuous Users Patients newly initiating Paliperidone Palmitate or on Paliperidone Palmitate at the time of enrollment
  Interventions: Drug: Paliperidone Palmitate -New and Continuous Users
- 004: Other Antipsychotics - New Starts Participants in the other antipsychotic cohort may be newly started on any oral or injectable antipsychotic other than Risperidone long acting injectable and Paliperidone Palmitate
  Interventions: Drug: Other Antipsychotics - New Starts

INTERVENTIONS:
Drug: Risperidone long acting injectable - New Starts — Patients who switch to Risperidone long acting injectable or receive an initial injection of Risperidone long acting injectable within the 30 days prior to enrollment will be eligible for inclusion in the Risperidone long acting injectable New Starts cohort.
  Groups: 001
Drug: Risperidone long acting injectable - Continuous Users — Patients who have been on Risperidone long acting injectable for at least 6 months before baseline, with no gaps between injections of more than 30 days will be eligible for inclusion in the Risperidone long acting injectable Continuous Users cohort.
  Groups: 002
Drug: Paliperidone Palmitate -New and Continuous Users — Patients newly initiating Paliperidone Palmitate or on Paliperidone Palmitate at the time of enrollment
  Groups: 003
Drug: Other Antipsychotics - New Starts — Participants in the other antipsychotic cohort may be newly started on any oral or injectable antipsychotic other than Risperidone long acting injectable and Paliperidone Palmitate
  Groups: 004

SUMMARY:
The purpose of this study is to build a data repository that can be used to understand pharmaceutical utilization patterns among patients being treated in community behavioral health organizations (CBHOs) for schizophrenia or bipolar I disorder.

DETAILED DESCRIPTION:
This is a prospective observational study of usual care of patients undergoing treatment for schizophrenia or bipolar I disorder at CBHOs. Up to 50 CBHOs will be selected as sites for this study. Treating clinicians at these sites will notify the designated research coordinators for this study when they are initiating a patient on a new antipsychotic medication (including risperidone long acting injectable or paliperidone palmitate) or if they are treating a patient with risperidone long acting injectable or paliperidone palmitate. New initiation will include patients not previously on any antipsychotic medication as well as those switched from one antipsychotic to another. Switches may include but are not limited to switches among different types of oral antipsychotics, from an oral antipsychotic to Long Acting Therapy (LAT), or from LAT to an oral antipsychotic. Site research staff will screen potential participants identified by the clinicians and enroll those meeting study criteria who consent to study participation. Sites will maintain a screening log of all potential participants. The target enrollment for this study is up to 2,450 participants. Enrollment by cohort will be monitored and sites will be notified to stop enrollment if target enrollment for a particular cohort has been reached. Eligible participants who consent to the study will be recruited into one of two samples: participants with a schizophrenia diagnosis (target n=2,250) and participants with a bipolar I disorder diagnosis (target n=200). There will be four cohorts: risperidone long acting injectable new starts (target n=475); risperidone long acting injectable continuous users (target n=75); paliperidone palmitate new starts or continuous users (target n=1,200); and other antipsychotic new starts (target n=700). During the entire study follow-up period participants will receive their medication per usual care in their treatment setting and no study drug will be provided. Enrolled participants will be followed prospectively over a 12-month study period, with interviews at baseline, 6 and 12 months. Sites will also abstract medical history and healthcare utilization information from the chart of each enrolled participant. There will be three chart abstractions (baseline, 6 Months, 12 Months). The baseline abstraction will cover services rendered in the 6 months prior to antipsychotic initiation or switch, or from their first visit to the CBHO if the individual did not receive services for as long as 6 months prior to initiation or switch. The 6M and 12M abstractions will each cover services rendered in the prior 6 months. When all three abstractions are complete, the data will cover the period from 6 months before baseline to 12 months after baseline. If a Serious Adverse Event (SAE) associated with a J&J medicinal product occurs the investigator will record it in the source document as well as fax the SAE form to J&J internal safety group within 24 hours. Treatment as usual

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia or bipolar I disorder
* Antipsychotic use in one of the following categories: Clinician ordered initiation of Risperidone long acting injectable in the 4 weeks prior to or on the day of enrollment (includes patients not previously on any antipsychotic medication and those switched from another antipsychotic)
* On continuous Risperidone long acting injectable for at least 6 months prior to enrollment (no gaps between injections>30 days)
* Clinician ordered initiation of Paliperidone Palmitate in the 4 weeks prior to or on the day of enrollment (includes patients not previously on any antipsychotic medication and those switched from another antipsychotic)
* or on continuous Paliperidone Palmitate for any time period prior to enrollment
* Clinician ordered initiation of another antipsychotic in the 4 weeks prior to or on the day of enrollment (includes patients not previously on any antipsychotic medication and those switched from another antipsychotic)
* Not enrolled in another clinical study
* Primary source of care for schizophrenia or bipolar I disorder is the recruiting CBHO
* Agrees to all study procedures/interviews
* must sign the study informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Currently participating in a clinical study (e.g. clinical trial or observational study) or participated in a clinical study within the past 30 days

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Potential participants will be identified by treating clinicians at the site. The study will enroll participants treated at participating sites for schizophrenia and bipolar I disorder. The study does not involve administration of a study drug, but will naturalistically follow partticipants in these medication cohorts at the time of enrollment: clinician ordered initiation or switch to LAT within past 4 weeks, clinician ordered initiation or switch to oral antipsychotic within past 4 weeks, continuous users ( greater than or equal to 6 months) of Risperdal long acting injectable, continuous users (greater than or equal to 1 month) of Invega Sustenna.
Sampling Method: Non-Probability Sample
Enrollment: 1066 (Actual)
Dates: Start 2010-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The number of psychiatric hospitalizations, non-psychiatric hospitalizations, emergency room visits, and CBHO visits. | Up to 12 months.

SECONDARY OUTCOMES:
Demographic and related participant information | Baseline, 6 and 12 months
The Structured Clinical Interview for Symptoms of Remission (SCI-SR) will be used to assess remission among participants with schizophrenia. | Baseline, 6 and 12 months
Quality of life will be measured using a modified version of the brief version of Lehman's Quality of Life Interview (QOLI). Developed specifically for use with persons with serious mental illness, and assesses satisfaction. | Baseline, 6 and 12 months
Psychiatric clinical characteristics will include the age first hospitalized for schizophrenia or bipolar I disorder (as applicable), or the years since first diagnosis. | Baseline, 6 and 12 months
The Personal and Social Performance Scale (PSP) will be used to measure functioning in four key areas: socially useful activities, including work and study; personal and social relationships; self -care; and disturbing behaviors. | Baseline, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (34):
- United States (34):
  - Neuropsychiatry Clinic and Research Center, Bullhead City, Arizona
  - Shanti Clinical Trials, Colton, California
  - Sun Valley Research Center, Imperial, California
  - South Coast Clinical Trials, Inc., Norwalk, California
  - Aurora Mental Health Center, Aurora, Colorado
  - LifeStream Behavioral Center, Inc., Leesburg, Florida
  - APF Research, Miami, Florida
  - River Edge Behavioral Health Center, Macon, Georgia
  - Human Service Center (Fayette Companies), Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Centerstone-Indiana Centerstone Research Institute, Bloomington, Indiana
  - Medical Development Centers LLC (Baton Rouge), Baton Rouge, Louisiana
  - Medical Development Centers LLC (Opelousas), Opelousas, Louisiana
  - OCCMHA/Community Network Services, Inc.: Oakland County Community Mental Health Authority, Farmington Hills, Michigan
  - Cherry Street Health Services, Grand Rapids, Michigan
  - Bootheel Counseling Services, Sikeston, Missouri
  - Burrell Behavioral Health, Springfield, Missouri
  - CenterPointe Institute of Research, St Louis, Missouri
  - Premier Psychiatric Research Institute, Lincoln, Nebraska
  - The Mental Health Center of Greater Manchester, Manchester, New Hampshire
  - Bergen Regional Medical Center, Paramus, New Jersey
  - St Joseph's Regional Medical Center, Paterson, New Jersey
  - Carolina Behavioral Care - Durham [CAREMARK], Durham, North Carolina
  - Carolina Behavioral Care - Henderson, Henderson, North Carolina
  - Carolina Behavioral Care - Hillsborough, Hillsborough, North Carolina
  - Lehigh Valley Hospital Dept. of Psychiatry, Allentown, Pennsylvania
  - Family Services of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Chestnut Ridge Counseling Services, Inc., Uniontown, Pennsylvania
  - South Shore Mental Health Center, Charleston, Rhode Island
  - Human Service Center (Fayette Companies), Pawtucket, Rhode Island
  - Centerstone-Tennessee Centerstone Research Institute, Nashville, Tennessee
  - Institute for Health Evaluation and Research Unlimited [IHEARU], Arlington, Texas
  - Center for Health Care Services, San Antonio, Texas
  - Frontier Institute-Research Department for Spokane Mental Health, Spokane, Washington

REFERENCES:
- [Derived] Joshi K, Mao L, Biondi DM, Millet R. The Research and Evaluation of Antipsychotic Treatment in Community Behavioral Health Organizations, Outcomes (REACH-OUT) study: real-world clinical practice in schizophrenia. BMC Psychiatry. 2018 Jan 29;18(1):24. doi: 10.1186/s12888-018-1594-1. PMID 29378547